CLINICAL TRIAL: NCT04281381
Title: A Prospective Analysis of Active Observation in Patients With Desmoid-Type Fibromatosis
Brief Title: Observing People With Desmoid-Type Fibromatosis
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 20-026
Record Dates: First submitted 2020-02-20; First posted 2020-02-24 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-03

CONDITIONS: Desmoid Fibromatosis
Keywords: Desmoid-Type Fibromatosis; Desmoid Fibromatosis; Desmoid; Fibromatosis; 20-026; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Desmoid Tumors; Fibroma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Desmoid Fibromatosis: Participants will have a clinical diagnosis of desmoid fibromatosis, either new or newly recurrent
  Interventions: Diagnostic Test: Cross-sectional imaging

INTERVENTIONS:
Diagnostic Test: Cross-sectional imaging — MRI with gadolinium contrast will be the imaging modality of choice. In patients with contraindications to MRI who instead undergo baseline evaluation by CT scan, tumor evaluation will be by serial CT scans with IV contrast throughout the study period.

SUMMARY:
The purpose of this study is to closely observe people with desmoid-type fibromatosis over 1 months.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of desmoid fibromatosis, either new or newly recurrent. Both patients with sporadic and FAP-associated disease will be eligible for inclusion. Patients with clinical diagnosis of desmoid (as assessed by MSK physician) but without pathologic diagnosis may be enrolled on the study to facilitate acquisition of appropriately protocoled baseline scans and allow for biospecimen collection; these patients will be replaced for purposes of analysis if pathology does not confirm clinical diagnosis.
* At least 18 years of age.
* Able to undergo cross-sectional imaging by either MRI or CT with intravenous contrast
* Disease detectable on cross-sectional imaging with target lesion measuring >/= 1 cm
* Eligible for management by active observation as assessed by primary MSK care provider
* Willing and able to sign an informed consent document

Exclusion Criteria:

* Symptomatic desmoid fibromatosis requiring narcotic pain control, resulting in intestinal fistulization, or requiring inpatient admission during the 3 months prior to enrollment
* Patients with intraabdominal desmoids greater than 7cm in diameter or localized within 1cm of the central mesenteric vessels and those with tumors in the head and neck
* KPS performance status </= 70 if performance status is limited due to tumor. Patients with low KPS performance status related to co-morbidities but without symptoms related to the tumor will be eligible for enrollment.
* Age less than 18 years old
* Strict contraindication for both cross-sectional MRI and CT imaging with intravenous contrast (e.g., as per standard institutional protocols regarding renal insufficiency or MRI incompatible implanted devices; patients requiring pre-medication to prevent contrast reactions will be eligible for study)
* Unable to grant reliable informed consent
* Ongoing systemic treatment for desmoid fibromatosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In most cases, patients will be identified by primary care providers in sarcoma medical and surgical oncology clinics.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-02-19 (Actual); Primary Completion 2026-02-19 (Estimated); Study Completion 2026-02-19 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 12 months
  The primary objective of this study is to estimate progression-free survival at 12 months, with the events defined by progression via radiographic criteria (RECIST 1.1).

CONTACTS AND LOCATIONS:
Overall Officials: Aimee M Crago, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org